CLINICAL TRIAL: NCT06118125
Title: Delay to Diagnosis and Management in Digestive Cancerology by the General Practitioner Within the City-hospital Network in the Context of Confinement Related to the Covid-19 Pandemic
Brief Title: Delay to Diagnosis in Digestive Cancerology by the General Practitioner Related to Covid-19 Pandemic Confinement
Status: Completed | Type: Observational
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Blanc-Bisson Christele, Doctor, University of Bordeaux
Other Study IDs: 2023-A02271-44
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Neoplasms, Colorectal; General Practitioner; Pandemic, COVID-19; Neoplasm, Liver; Neoplasms Pancreatic; Diagnosis; Advanced Cancer
Keywords: digestive cancer, covid
MeSH Terms: conditions — Colorectal Neoplasms; COVID-19; Liver Neoplasms; Pancreatic Neoplasms; Disease; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2019: patients diagnosed in 2019
- 2020: patients diagnosed in 2020

SUMMARY:
Objective: the pre-hospital management of cancers is little known in General Medicine. The first lockdown related to the COVID-19 pandemic led to the closure of health facilities. Investigators were interested in the diagnosis and care pathway of digestive cancers in post-confinement in General Medicine in Nouvelle-Aquitaine.

DETAILED DESCRIPTION:
Method: patient records discussed in Digestive Oncology CPR of Bordeaux University Hospital for the first time from June 1 to August 31, 2020 and over the same period in 2019 were included. A questionnaire on the dates of the first symptoms, first consultation with the general practitioner, imaging examination and access to the specialist was sent to the general practitioner. The primary outcome was time from onset to date of first MDT.

ELIGIBILITY:
Inclusion Criteria:

* residing in New Aquitaine and
* whose general practitioner practiced in New Aquitaine
* malignant tumors of the esophagus, stomach, small intestine, colon, recto-sigmoid junction, rectum, anus and anal canal, liver and intrahepatic bile ducts, extrahepatic bile ducts, gallbladder and pancreas.
* to have had at least one consultation or hospitalization in the digestive pole of the Bordeaux University Hospital within 6 months after the MDT.

Exclusion Criteria:

* Patients under 18 years of age,
* who had already had a MDT for this cancer,
* whose date of first MDT was outside the inclusion dates,
* whose new cancer was a digestive metastasis of a primary of another location,
* who did not have French health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female under 18 years old
  * residing in New Aquitaine and
  * whose general practitioner practiced in New Aquitaine
  * malignant tumors of the esophagus, stomach, small intestine, colon, recto-sigmoid junction, rectum, anus and anal canal, liver and intrahepatic bile ducts, extrahepatic bile ducts, gallbladder and pancreas.
  * to have had at least one consultation or hospitalization in the digestive pole of the Bordeaux University Hospital within 6 months after the MDT.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
time from date of first symptoms of cancer to the date of first MDT | DAYS
  time from date of first symptoms of cancer to the date of first MDT

SECONDARY OUTCOMES:
time from date of first symptoms to date of first consultation with a general practitioner, | DAYS
  time from date of first symptoms to date of first consultation with a general practitioner,
time from date of first symptoms to first imaging or specific examination, | DAYS
  difficulties in referral to imaging,
time from date of first symptoms to consultation with a specialist, | DAYS
  difficulties in referral to a specialist,
stage of pathology by type of cancer, | at inclusion
  stage of pathology by type of cancer according to TNM classification (tumor, node, metastatic status)
frequency of different types of cancer, | at inclusion
  PERCENTAGE of each type of cancers in this study
overall survival. | MONTHS, time from from date of first symptoms to date of death
  overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Blanc-Bisson Christele, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No